CLINICAL TRIAL: NCT01144780
Title: Investigation of Dysregulated Signaling in Myeloproliferative Disorders Via Multiparameter Phospho-specific Flow Cytometry
Brief Title: Investigation of Dysregulated Signaling in MPD Via Multiparameter Phospho-specific Flow Cytometry
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-14723; HEMMPD0011 (Other: OnCore); SU-07092009-3060 (Other: Stanford)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Myeloproliferative Disorders; Myeloproliferative Disorders (MPD)
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and bone marrow
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to better understand the underlying pathogenetic mechanisms of myeloproliferative disorders (MPDs). We will collect peripheral blood samples from MPD patients and utilize multiparameter phospho-specific flow cytometry to investigate dysregulated signaling in blood cells from these patients. This will provide deeper insights into the pathogenesis of MPDs and may lead to the identification of novel targets for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:Any patient who carries a diagnosis of a myeloproliferative disorder (MPD). Exclusion Criteria:Any patient who is not willing to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who carries a diagnosis of a myeloproliferative disorder (MPD).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robert Gotlib, Principal Investigator — Stanford University; Stephen Tracy Oh, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States